CLINICAL TRIAL: NCT05416996
Title: Feasibility Study of Randomizing Patients to Telemedicine Shared Medical Appointments Versus Telemedicine Single Visits for Men With Prostate Cancer on Active Surveillance
Brief Title: A Study of Telemedicine Shared Medical Appointments (SMAs) Versus Individual Telemedicine Visits for People With Prostate Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-184
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Telemedicine; Shared Medical Appointments; Individual Telemedicine Visits; 22-184
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shared Medical Appointments
- Usual Care Appointments

SUMMARY:
The purpose of this study is to see if a telemedicine group doctor's appointment is a practical (feasible) and acceptable method for following people with prostate cancer being managed with active surveillance when compared with the usual approach of individual telemedicine visits, which involve the participant visiting a doctor on their own. The researchers will compare the telemedicine group and individual visits by measuring on participant satisfaction and quality of life in each type of visit. Telemedicine is the use of secure video technology on a desktop computer, laptop, smartphone, or tablet to provide and receive healthcare from a distance.

ELIGIBILITY:
Inclusion Criteria:

* A scheduled appointment for a subsequent Active Surveillance (AS) follow-up visit for management of localized prostate cancer
* Biopsy Gleason score 3+3=6 (Grade Group 1) or biopsy Gleason score 3+4=7 (Grade Group 2)
* Clinical T stage ≤T2B
* Access to a device with Zoom
* Ability to speak and understand English

Exclusion Criteria:

* Plan to undergo a prostate biopsy at this follow-up visit

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer
Study Population: Patients will be recruited through two routes: 1) by physician invitation during routine Active Surveillance (AS) office visits or 2) by the physician's assistant or research team calling.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
accrual number | 1 year
patient satisfaction | 1 week
  using MSK Engage portal survey

SECONDARY OUTCOMES:
adherence to active surveillance | 6 months
  the number who drop out of AS in the absence of disease progression

OTHER OUTCOMES:
Functional status | 1 year
  These patient-reported outcomes are captured electronically and using validated questionnaires as part of the standard of care at MSK via MSK Engage. (anxiety, quality of life, urinary function, and erectile function)

CONTACTS AND LOCATIONS:
Overall Officials: Behfar Ehdaie, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm